CLINICAL TRIAL: NCT04182451
Title: A Multi-center, Prospective Clinical Trial Evaluating the Effect of Meso Wound Matrix in the Treatment of Chronic Non-healing Diabetic Foot Ulcers (DFUs).
Brief Title: Effect of Meso Wound Matrix in the Treatment of DFUs
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: SerenaGroup, Inc. (Network)
Collaborators: DSM Biomedical, Inc. (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MESO-001
Record Dates: First submitted 2019-11-27; First posted 2019-12-02 (Actual); Last update posted 2023-04-26 (Actual); Status verified 2023-04

CONDITIONS: Diabetic Foot Ulcers (DFUs)
Keywords: Chronic wounds
MeSH Terms: conditions — Diabetic Foot

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- Meso Wound Matrix and Standard of Care (Experimental): This is a single arm study
  Interventions: Device: Meso Wound Matrix

INTERVENTIONS:
Device: Meso Wound Matrix — Subjects who meet eligibility criteria will receive standard of care and Meso Wound Matrix.
  The standard of care therapy in this study is offloading of the DFU, appropriate sharp or surgical debridement, and aggressive infection management with the use of appropriate dressings. Total contact casting or fixed ankle walker will be used for off-loading. Wound Matrix is an acellular scaffold to reinforce and repair soft tissue defects. Subjects may receive up to eight applications of Meso Wound Matrix. Subjects whose study ulcer does not heal after eight applications will receive only SOC treatment for 4 additional weeks.

SUMMARY:
This is a prospective trial designed to evaluate the use of Meso Wound Matrix (DSM Biomedical, Exton, PA) in Wagner grade 1 and 2 DFUs.

DETAILED DESCRIPTION:
At the Screening Visit (SV), written informed consent will be obtained from the subject by the Investigator or designee before the performance of any other protocol-specific procedure. The Investigator will select the Index (study) ulcer. Each subject will have only one DFU selected as the Index (study) ulcer. If the subject has more than one ulcer at the SV, the Investigator will select the largest ulcer that meets the eligibility criteria of the protocol as the Index (study) ulcer.The SV is designed to determine whether subjects are eligible to proceed to the Treatment Phase of the study. Those subjects who meet the eligibility criteria will transition to Treatment Visit 1 (TV1) on the same day as the SV.

Subjects who meet eligibility criteria at the SV will receive Meso Wound Matrix (DSM Biomedical, Exton, PA) and standard of care. During the Treatment Phase, subjects will be evaluated on a weekly basis. Efficacy evaluations each week will include Investigator assessment of ulcer healing and measurements of ulcer size using digital photographic planimetry. Safety evaluations during the Treatment Phase will consist of adverse event assessments at each visit. Subjects may receive up to eight applications of Meso Wound Matrix. Subjects whose study ulcer does not heal after eight applications will receive only SOC treatment for 4 additional weeks. Subjects whose ulcers do not achieve closure at or by 12 weeks or who experience an amputation will be deemed treatment failures.

ELIGIBILITY:
Inclusion Criteria:

1. At least 18 years old
2. Presence of a diabetic foot ulcer, Wagner 1 or 2 grade, extending at least through the dermis or subcutaneous tissue and may involve the tendon or muscle provided it is below the medial aspect of the malleolus
3. The index ulcer will be the largest ulcer if 2 or more ulcers are present on the same extremity. If other ulcerations are present on the same foot they must be more than 2 cm apart from the index ulcer.
4. Index ulcer (i.e. current episode of ulceration) has been present for greater than 4 weeks prior to the initial screening visit
5. Study ulcer size is a minimum of 0.75 cm2 and a maximum of 5 cm2 at first treatment visit
6. Adequate circulation to the affected extremity as demonstrated by a transcutaneous oxygen measurement (TCOM) or a skin perfusion pressure (SPP) measurement of ≥ 30 mmHg, or an Ankle Brachial Index (ABI - measure of blood flow to the ankle) between 0.7 and ≤ 1.3
7. Females of childbearing potential must be willing to use acceptable methods of contraception (birth control pills, barriers, or abstinence)
8. Subject understands and is willing to participate in the clinical study and can comply with weekly visits and the follow-up regimen
9. Subject has read and signed the IRB approved Informed Consent Form before screening procedures are undertaken
10. The subject is willing to apply a porcine based product to the wound

Exclusion Criteria:

1. Study ulcer(s) deemed by the investigator to be caused by a medical condition other than diabetes.
2. Index ulcer, in the opinion of the investigator, is suspicious for cancer and should undergo an ulcer biopsy to rule out a carcinoma of the ulcer.
3. Subjects with a history of more than two weeks treatment with immunosuppressants (including systemic corticosteroids >10mg daily dose), cytotoxic chemotherapy, or application of topical steroids to the ulcer surface within one month prior to first Screening Visit, or who receive such medications during the screening period, or who are anticipated to require such medications during the course of the study.
4. History of radiation at the ulcer site.
5. Presence of any condition(s) which seriously compromises the subject's ability to complete this study or has a known history of poor adherence with medical treatment.
6. Osteomyelitis or bone infection of the affected foot or leg as verified by X-ray within 30 days prior to Randomization.
7. Subject is pregnant or breast-feeding.
8. The study ulcer with a history of treatment with hyperbaric oxygen of cellular or Tissue-based Product (CTP) within 30 days of randomization.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2019-12-05 (Actual); Primary Completion 2022-05-17 (Actual); Study Completion 2023-03-01 (Actual)

PRIMARY OUTCOMES:
Efficacy of Meso Wound Matrix | 12 Weeks
  Efficacy of Meso Wound Matrix as an adjunctive treatment in facilitating wound healing in Wagner 1 and 2 grade DFUs when compared to traditional and well-established controls.

SECONDARY OUTCOMES:
Wound Surface Area Reduction | 4 Weeks
  Proportion of wounds with surface area reduction of greater than 40% at 4 weeks
Wound Closure | 12 Weeks
  Proportion of wounds healed at 12 weeks
Adverse Events | 12 Weeks
  Incidence of adverse events
Device Utilization | 12 Weeks
  Graft wastage
Health Economics | 12 Weeks
  Cost to heal

CONTACTS AND LOCATIONS:
Locations (3):
- United States (3):
  - Royal Research, Pembroke Pines, Florida
  - Foot & Ankle Wellness Clinic, Ford City, Pennsylvania
  - D&P Medical Group, Pittsburgh, Pennsylvania